CLINICAL TRIAL: NCT01057459
Title: Natural Killer Cell KIR and HLA Genotypes May Predict Response to Antibody Therapy in Follicular Lymphoma
Brief Title: DNA Analysis in Predicting Response to Antibody Therapy in Patients With Follicular Lymphoma Treated on Clinical Trials CALGB-50402 or CALGB-50701
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150905; CDR0000664103; NCI-2011-02204 (Registry Identifier: NCI Physician Data Query); U10CA180821 (NIH)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Lymphoma
Keywords: Stage II Grade 1 Contiguous Follicular Lymphoma; Stage II Grade 1 Non-Contiguous Follicular Lymphoma; Stage II Grade 2 Contiguous Follicular Lymphoma; Stage II Grade 2 Non-Contiguous Follicular Lymphoma; Stage II Grade 3 Contiguous Follicular Lymphoma; Stage II Grade 3 Non-Contiguous Follicular Lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (biomarkers and treatment outcomes): Genomic DNA is extracted from previously collected blood samples for KIR and HLA genotyping and polymorphism analysis.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies deoxyribonucleic acid (DNA) analysis in predicting response to antibody therapy in patients with follicular lymphoma treated on clinical trials Cancer and Leukemia Group B (CALGB)-50402 or CALGB-50701. Studying samples of blood from patients with follicular lymphoma in the laboratory may help doctors predict how well patients will respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To test the hypothesis that killer immunoglobulin-like receptor (KIR) and human leukocyte antigen (HLA) genotypes predict overall response (partial response [PR], complete response[CR], and unconfirmed complete response [CRu]) within 12 months to rituximab-containing monoclonal antibody combinations in follicular lymphoma patients treated on CALGB protocols 50402 and 50701.

SECONDARY OBJECTIVES:

I. To test the hypothesis that KIR and HLA genotypes are associated with survival outcomes (progression-free survival [PFS] and overall survival [OS]) in follicular lymphoma patients treated with rituximab-containing monoclonal antibody combinations on CALGB protocols 50402 and 50701.

OUTLINE:

Genomic DNA is extracted from previously collected blood samples for KIR and HLA genotyping and polymorphism analysis.

ELIGIBILITY:
Inclusion Criteria:

* Untreated follicular lymphoma
* Has received rituximab-containing monoclonal antibody therapy on CALGB-50402 or CALGB-50701
* Patients have previously provided informed consent allowing correlative studies on genomic DNA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with follicular lymphoma treated on CALGB 50402 or 50701 protocols
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2014-06-23 (Actual); Study Completion 2014-06-23 (Actual)

PRIMARY OUTCOMES:
overall response | Baseline

SECONDARY OUTCOMES:
Progression-free survival | Baseline
Overall survival | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Venstrom, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States